CLINICAL TRIAL: NCT07216508
Title: Post-discharge Glycemic Control After Liver Transplant and Impact on Transplant Outcomes
Brief Title: Liver Transplant CGM
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Grenye O'Malley, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-24-01098
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Liver Transplant; Post Transplant Diabetes; Type 2 Diabetes
Keywords: liver transplant; hyperglycemia; diabetes; continuous glucose monitoring; glucose sensor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Participants post liver transplant: Participants who are discharged from after liver transplant.
  Interventions: Device: Libre 3+

INTERVENTIONS:
Device: Libre 3+ — Blinded CGM will be worn by all participants
  Other Names: blinded CGM

SUMMARY:
This investigator initiated study aims to describe continuous glucose monitoring (CGM) based glycemic metrics after discharge from liver transplant and assess relationship with glycemic metrics and liver transplant outcomes.

DETAILED DESCRIPTION:
Liver transplant participants will be recruited. Participants will wear a blinded sensor after hospital discharge for up to 30 days. Data can be shared with participant and the providers retrospectively. Participants will be invited to wear another blinded sensor at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

• inpatient liver transplant participants who have had an inpatient glucose greater than 180mg/dL

Exclusion Criteria:

* having a planned discharge to a rehabilitation or nursing facility,
* a contraindication to sensor placement,
* if discharge is anticipated to be >30 days post-transplant, or
* if recent transplant also included a kidney or pancreas transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inpatient liver transplant participants who have had an inpatient glucose greater than 180mg/dL
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2027-10-05 (Estimated)

PRIMARY OUTCOMES:
Time in range | 28 days
  Time in range 70-180mg/dL

SECONDARY OUTCOMES:
Percent time >180mg/dL | 28 days
  Percent time >180mg/dL
Percent time >250mg/dL | 28 days
  Percent time >250mg/dL
Percent time <70mg/dL | 28 days
  Percent time <70mg/dL
Percent time <54mg/dL | 28 days
  Percent time <54mg/dL
Transplant outcomes | 1 year
  Rate and time to of wound complications, vascular complications, biliary complications, acute kidney injury, transplant rejection, and readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Grenye O'Malley, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Identifying dates